CLINICAL TRIAL: NCT01601054
Title: Supplemental Anterior Lumbar Interbody Fusion in Posterior Instrumented Fusion in Surgical Treatment of Spinal Deformities. A Randomized Study
Brief Title: Supplemental Anterior Lumbar Interbody Fusion (ALIF) in Spinal Deformity
Acronym: SALIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Benny Dahl, MD, PhD, Professor of Spine Surgery, Rigshospitalet, Denmark
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-2-2012-003
Record Dates: First submitted 2012-05-14; First posted 2012-05-17 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Spinal Deformity
Keywords: spine; deformity; instrumentation; ALIF
MeSH Terms: conditions — Congenital Abnormalities | interventions — Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior lumbar interbody fusion (Active Comparator): Anterior lumbar interbody fusion using a tantalum cage. Cage will be inserted through a left sided retroperitoneal approach.
  Interventions: Device: Tantalum cage from Zimmer
- Posterior instrumentation alone (Active Comparator): Posterior pedicle screw instrumentation
  Interventions: Device: Tantalum cage from Zimmer

INTERVENTIONS:
Device: Tantalum cage from Zimmer — A tantalum cage will be inserted through a left sided retroperitoneal approach
  Other Names: Tantalum

SUMMARY:
Within the last decade there has been an increase in the number of surgical procedures for deformities of the spine. This is caused by the increase in the elderly population, improved surgical techniques and an increased number of patients who have undergone previous surgical treatment for degenerative conditions of the spine. Surgical treatment of spinal deformities bears a revision rate between 15 and 30% depending on definition, and one of the primary reasons for revision surgery is implant loosening in the lumbosacral region.

The hypothesis of the study is that a procedure resulting in anterior fusion of the lumbar spine in addition to the usual posterior instrumentation can reduce the revision rate with 50%.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more of age
* planned posterior instrumented fusion from thoracic spine to sacrum and/or ilium

Exclusion Criteria:

* malignancy
* infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Revision | 12 months
  Surgical revision rate because of implant failure or pseudarthrosis within 12 months after primary procedure

CONTACTS AND LOCATIONS:
Overall Officials: Benny Dahl, MD, Principal Investigator — University of Copenhagen, Rigshospitalet
Locations (1):
- Spine Unit, Rigshospitalet, 9 Blegdamsvej, Copenhagen, Osterbro, Denmark